CLINICAL TRIAL: NCT01957176
Title: Study 200170: A Rollover Study to Provide Continued Treatment With Eltrombopag
Brief Title: A Rollover Study to Provide Continued Treatment With Eltrombopag
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200170; 2013-001371-20 (EudraCT Number); CETB115A2X01B (Other: Novartis)
Record Dates: First submitted 2013-10-04; First posted 2013-10-08 (Estimated); Results first posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-11

CONDITIONS: Thrombocytopaenia
Keywords: myelodysplastic syndromes; thrombocytopenia; acute myeloid leukemia; idiopathic thrombocytopenic purpura; Eltrombopag; pediatrics
MeSH Terms: conditions — Thrombocytopenia; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Purpura, Thrombocytopenic, Idiopathic | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A (Myelodysplastic syndrome (MDS)/ Acute myeloid leukemia (AML) adult subjects) (Experimental): All subjects in this cohort received eltrombopag (ELT) at the dose that they were receiving at the time of the transition visit, except in the case where the subject required a dose modification. The range of doses of ELT that were used in this cohort were from 50 to 300 mg once daily (OD) for subjects of non-East Asian heritage. The dose ranges for subjects of East Asian heritage (i.e., Japanese, Chinese, Taiwanese, Thai and Korean) were 25 to 150 mg. Dose adjustments (if required) were done depending on each subject's platelet counts.
  Interventions: Drug: Eltrombopag (ELT)
- Cohort B (Idiopathic thrombocytopenic purpura (ITP) adult subjects) (Experimental): All subjects in this cohort received ELT at the dose that they were receiving at the time of the transition visit, except in the case where the subject required a dose modification. The range of doses of ELT that were used in this cohort were from 12.5 to 75 mg. Dose adjustments (if required) were done depending on each subject's platelet counts.
  Interventions: Drug: Eltrombopag (ELT)
- Cohort C (Idiopathic thrombocytopenic purpura (ITP) pediatric subjects) (Experimental): All subjects in this cohort received ELT at the dose that they were receiving at the time of the transition visit, except in the case where the subject required a dose modification. The range of doses of ELT that were used in this cohort were from 12.5 to 75 mg. Dose adjustments (if required) were done depending on each subject's platelet counts.
  Interventions: Drug: Eltrombopag (ELT)

INTERVENTIONS:
Drug: Eltrombopag (ELT) — Subjects were dosed with ELT tablets or powder for oral suspension (PfOS) based on the dosage form used in the parent study. ELT tablets were white, round film coated tablets containing ELT olamine equivalent to 12.5 mg, 25 mg, 50 mg, 75 mg and 100 mg of ELT. ELT PfOS was a reddish-brown to yellow powder contained inside an elongated sachet. Each sachet contained ELT olamine equivalent to 20 mg of ELT per gram of powder.
  Other Names: SB-497115

SUMMARY:
The objective of this study was to provide continued treatment with eltrombopag for subjects who were participating in a Novartis-sponsored investigational study with eltrombopag (parent studies 114968/ASPIRE (NCT01440374), PMA112509 (NCT00903422), and TRA105325/EXTEND (NCT00351468), receiving clinical benefit without unacceptable toxicity and to collect long-term safety data.

DETAILED DESCRIPTION:
This Phase IV, multicenter, non-randomized, open-label, uncontrolled, rollover study was designed to provide continued access to eltrombopag to eligible subjects. As this study was a rollover study, the subjects were enrolled into this study from the parent studies.

There were 3 cohorts in this study:

Cohort A: Adult subjects who have completed study treatment with eltrombopag during their participation in a parent study for MDS/AML (i.e., 114968/ASPIRE and PMA112509).

Cohort B: Adult subjects who have completed study treatment with eltrombopag during their participation in a parent study for ITP (i.e., TRA105325/EXTEND).

Cohort C: Pediatric subjects who have completed study treatment with eltrombopag during their participation in a parent study for ITP. Once a subject turned 18 years of age, they might remain in the study and follow the Cohort B procedures. No pediatric subjects were enrolled in this cohort/study.

The study consisted of a transition visit, study treatment visits, and a follow-up visit. Subjects in Cohort A and Cohort B completed the Transition visit assessments and then returned for their next schedule visit as per the Visit schedule. In the study treatment visit, subjects received a starting dose of eltrombopag at the same dose and administration that they were receiving at the time of their last study treatment visit in the parent study.

Safety was evaluated through physical examinations, clinical laboratory tests, and monitoring of adverse events. Additional safety assessments were done as per standard of care and/or when medically indicated.

Assessment of clinical benefit was performed throughout the study using local standard of care as determined by the Investigator to determine continued study participation and treatment with eltrombopag. Only subjects considered by the Investigator to be receiving clinical benefit without unacceptable toxicity may continue on study treatment. Once treatment with eltrombopag was permanently discontinued, the subject would attend the follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent has been obtained from the subject (or subject's legally acceptable representative) prior to performance of any study-specific procedure.
* The subject is participating in a GSK sponsored investigational study of eltrombopag (parent study) within the past 28 days and is receiving clinical benefit without unacceptable toxicity as determined by the investigator.
* Subjects with a QTc <450 millisecond (msec) or <480 msec for subjects with bundle branch block. The QTc is the QT interval corrected for heart rate according to either Bazett's formula (QTcB), Fridericia's formula (QTcF) or another method, machine or manual overread. For subject eligibility and withdrawal QTcF will be used. For purposes of data analysis, QTcF will be used. The QTc should be based on single or averaged QTc values of triplicate electrocardiograms (ECGs) obtained over a brief recording period.
* Women must be either of non-child bearing potential or women with child-bearing potential and men with reproductive potential must be willing to practice acceptable methods of birth control during the study.
* Women of childbearing potential must have a negative serum pregnancy test within 14 days of the first dose of study treatment and agree to use effective contraception, during the study and for 4 weeks following the last dose of study treatment.
* Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception from time of first dose until 16 weeks after the last dose of study treatment.
* In France, a subject will be eligible for inclusion in this study only if either affiliated to, or a beneficiary of, a social security category.

Exclusion Criteria:

* Permanent discontinuation of eltrombopag in the parent study based upon the study treatment discontinuation or study withdrawal criteria from the parent study. Subjects who permanently discontinued treatment because they completed all study related treatments remain eligible.
* The subject is pregnant or a lactating female.
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions at the time of transition to this study that could interfere with subject's safety, obtaining informed consent or compliance with the study procedures, in the opinion of the investigator or GSK Medical Monitor.
* French subjects: The French subject has participated in any study using an investigational drug during the previous 30 days, with the exception of eltrombopag, in the parent study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-10-15 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- Novartis Investigative Site, Leuven, Belgium
- Novartis Investigative Site, Shanghai, China
- Novartis Investigative Site, Paris, France
- Greece (2):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Heraklion, Crete
- Novartis Investigative Site, Shatin, Hong Kong
- Novartis Investigative Site, Tullamore, Ireland
- Novartis Investigative Site, Amsterdam, Netherlands
- Novartis Investigative Site, San Isidro, Lima region, Peru
- Novartis Investigative Site, Chorzów, Poland
- Novartis Investigative Site, Bucharest, Romania
- Novartis Investigative Site, Seoul, South Korea
- Novartis Investigative Site, Sousse, Tunisia

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 22 subjects were enrolled in 14 centers in 12 countries (Belgium, China, France, Greece, Hong Kong, Ireland, Korea, Republic of., Netherlands, Peru, Poland, Romania, Tunisia).
Period: Overall Study
Arm/Group | Cohort A (Myelodysplastic Syndrome (MDS)/ Acute Myeloid Leukemia (AML) Adult Subjects) | Cohort B (Idiopathic Thrombocytopenic Purpura (ITP) Adult Subjects)
Started (All the subjects who were treated with at least one dose of eltrombopag were included in the All Treated Subjects analysis set (ATS analysis set)) | 8 | 14
Completed | 3 | 13
Not Completed | 5 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Physician Decision | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A (Myelodysplastic Syndrome (MDS)/ Acute Myeloid Leukemia (AML) Adult Subjects) | Cohort B (Idiopathic Thrombocytopenic Purpura (ITP) Adult Subjects) | Total
Number analyzed (Participants) | 8 | 14 | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.8 (7.57) | 59.5 (13.18) | 64.7 (13.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 12 | 15
  Male | 5 | 2 | 7
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaskan Native | 0 | 2 | 2
  Asian - East Asian Heritage | 1 | 5 | 6
  White - Arabic/North African Heritage | 0 | 6 | 6
  White - White/Caucasian/European Heritage | 7 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: The distribution of adverse events was done via the analysis of frequencies for Adverse Events (AEs) and Serious Adverse Events (SAEs), through the monitoring of relevant clinical and laboratory safety parameters. Only descriptive analysis performed.
Time Frame: From the time of transition visit until 30 days after last dose of study treatment, assessed up to approximately 100 months.
Population: All treated subjects (ATS): All subjects who received at least one dose of eltrombopag on this study were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Myelodysplastic Syndrome (MDS)/ Acute Myeloid Leukemia (AML) Adult Subjects) | Cohort B (Idiopathic Thrombocytopenic Purpura (ITP) Adult Subjects)
Number analyzed (Participants) | 8 | 14
Participants
  Adverse Events (AEs) | 7 | 12
  Serious Adverse Events (SAEs) | 6 | 7

ADVERSE EVENTS:
Time Frame: From the time of transition visit until 30 days after last dose of study treatment, assessed up to approximately 100 months.
Description: Any sign or symptom that occurs during the treatment period plus 30 days post-treatment.
Groups:
- All Subjects: All enrolled subjects in the study
Arm/Group | Cohort A (Myelodysplastic Syndrome (MDS)/ Acute Myeloid Leukemia (AML) Adult Subjects) | Cohort B (Idiopathic Thrombocytopenic Purpura (ITP) Adult Subjects) | All Subjects
All-Cause Mortality (participants affected / at risk) | 3/8 | 2/14 | 5/22
Serious Adverse Events (participants affected / at risk) | 6/8 | 7/14 | 13/22
Other Adverse Events (participants affected / at risk) | 7/8 | 12/14 | 19/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (Myelodysplastic Syndrome (MDS)/ Acute Myeloid Leukemia (AML) Adult Subjects) (N=8) | Cohort B (Idiopathic Thrombocytopenic Purpura (ITP) Adult Subjects) (N=14) | All Subjects (N=22)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 1
Encephalitis (Infections and infestations) | 0 | 1 | 1
Encephalitis viral (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 2
Sepsis (Infections and infestations) | 2 | 0 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1 | 1
Subdural hygroma (Nervous system disorders) | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (Myelodysplastic Syndrome (MDS)/ Acute Myeloid Leukemia (AML) Adult Subjects) (N=8) | Cohort B (Idiopathic Thrombocytopenic Purpura (ITP) Adult Subjects) (N=14) | All Subjects (N=22)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 4
Eosinophilia (Blood and lymphatic system disorders) | 0 | 5 | 5
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 3 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 1
Monocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Neutrophilia (Blood and lymphatic system disorders) | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 2
Tachycardia (Cardiac disorders) | 0 | 2 | 2
Cataract (Eye disorders) | 0 | 1 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 1
Diabetic retinopathy (Eye disorders) | 0 | 1 | 1
Ocular hyperaemia (Eye disorders) | 0 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 5
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 | 1 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 2 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Asthenia (General disorders) | 1 | 2 | 3
Chest pain (General disorders) | 1 | 0 | 1
Chills (General disorders) | 1 | 0 | 1
Discomfort (General disorders) | 0 | 1 | 1
Face oedema (General disorders) | 0 | 1 | 1
Fatigue (General disorders) | 2 | 0 | 2
Inflammation (General disorders) | 1 | 0 | 1
Mucosal haemorrhage (General disorders) | 0 | 1 | 1
Oedema peripheral (General disorders) | 3 | 1 | 4
Pyrexia (General disorders) | 4 | 3 | 7
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0 | 1
Ocular icterus (Hepatobiliary disorders) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1
COVID-19 (Infections and infestations) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 1
Conjunctivitis (Infections and infestations) | 0 | 1 | 1
Ear infection (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 3 | 3
Genital infection (Infections and infestations) | 0 | 1 | 1
Gingivitis (Infections and infestations) | 0 | 2 | 2
Herpes zoster (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 1 | 3 | 4
Kidney infection (Infections and infestations) | 0 | 1 | 1
Lip infection (Infections and infestations) | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 2 | 2
Onychomycosis (Infections and infestations) | 0 | 1 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 1
Paronychia (Infections and infestations) | 0 | 1 | 1
Periodontitis (Infections and infestations) | 0 | 1 | 1
Pharyngotonsillitis (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 2
Respiratory tract infection (Infections and infestations) | 1 | 1 | 2
Rhinitis (Infections and infestations) | 0 | 1 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1 | 1
Tooth infection (Infections and infestations) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 5 | 6
Urinary tract infection (Infections and infestations) | 0 | 3 | 3
Vaginal infection (Infections and infestations) | 0 | 1 | 1
Viral infection (Infections and infestations) | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Scratch (Injury, poisoning and procedural complications) | 1 | 0 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 2 | 2
Alanine aminotransferase increased (Investigations) | 1 | 3 | 4
Apolipoprotein E abnormal (Investigations) | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 3 | 4
Blood albumin decreased (Investigations) | 0 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 3 | 3
Blood glucose increased (Investigations) | 0 | 1 | 1
Blood pressure increased (Investigations) | 0 | 1 | 1
Blood urea increased (Investigations) | 0 | 2 | 2
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 1
Globulins increased (Investigations) | 0 | 1 | 1
Haematocrit increased (Investigations) | 0 | 1 | 1
Haemoglobin decreased (Investigations) | 1 | 0 | 1
Haemoglobin increased (Investigations) | 0 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 1
Neutrophil count increased (Investigations) | 0 | 2 | 2
Platelet count increased (Investigations) | 0 | 2 | 2
Protein total increased (Investigations) | 0 | 1 | 1
Urinary occult blood positive (Investigations) | 0 | 1 | 1
Urine ketone body present (Investigations) | 0 | 1 | 1
Weight decreased (Investigations) | 1 | 0 | 1
White blood cell count increased (Investigations) | 2 | 2 | 4
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 2
Headache (Nervous system disorders) | 1 | 5 | 6
Lethargy (Nervous system disorders) | 1 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 2 | 2
Nocturia (Renal and urinary disorders) | 1 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 1
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 2 | 2
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 1
Scrotal oedema (Reproductive system and breast disorders) | 1 | 0 | 1
Bronchial irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Haematoma (Vascular disorders) | 1 | 1 | 2
Hot flush (Vascular disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 4 | 5
Hypertensive crisis (Vascular disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-04-06): https://cdn.clinicaltrials.gov/large-docs/76/NCT01957176/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/76/NCT01957176/SAP_001.pdf